CLINICAL TRIAL: NCT03825965
Title: The Effect of Cannabinoids vs. Placebo on Persistent Post-surgical Pain Following Total Knee Arthroplasty: A Multicenter, Randomized Pilot Trial
Brief Title: Cannabinoids vs. Placebo on Persistent Post-surgical Pain Following TKA: A Pilot RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cannabis TKA Pilot Trial
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee arthroplasty; Cannabis; Pilot trial; Persistent post-surgical pain
MeSH Terms: conditions — Osteoarthritis, Knee; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPL-001 (CBD: THC 25:1) (Experimental): 125mg CBD/5 mg THC oil for oral use
  Interventions: Drug: MPL-001 (CBD: THC 25:1)
- Placebo (Placebo Comparator): Visually identical placebo (medium chain triglyceride oil)
  Interventions: Drug: Placebo oil for oral use

INTERVENTIONS:
Drug: MPL-001 (CBD: THC 25:1) — 25:1 cannabidiol (CBD): tetrahydrocannabinol (THC) oral formulation, with a concentration of 50 mg/mL CBD and 2 mg/mL THC, oil- Liquid for oral use
  Arms: MPL-001 (CBD: THC 25:1)
Drug: Placebo oil for oral use — Placebo is Medium-chain triglycerides oil with identical features (in appearance, flavour, and odour) to the MPL-001 oil.
  Arms: Placebo

SUMMARY:
Each year, approximately 75,000 Canadians undergo knee replacement surgery, and up to 25% develop persistent post-surgical pain. Persistent post-surgical pain is associated with depression, anxiety, unemployment, and reduced quality of life. Chronic pain after surgery is often managed with opioid therapy, which typically provides only modest benefits and is associated with rare but serious adverse events, such as overdose and death. A number of studies have found that greater pain just before and after knee replacement surgery is associated with the development of chronic pain, suggesting that reducing peri-operative pain may help prevent persistent post-surgical pain.

Medicinal cannabis has begun to emerge as a potential therapy for pain reduction, and produces effects largely due to 2 active components: (1) cannabidiol (CBD), and (2) tetrahydrocannabinol (THC). Studies of CBD have shown analgesic, anti-inflammatory, and anti-anxiety properties, but without the psychoactive effects (feeling 'high') that THC produces. This study will assess the feasibility of a definitive trial to explore whether adding CBD dominant vs. placebo to usual care before and after surgery can reduce the rate of persistent post-surgical pain after total knee replacement. This study will randomize 40 patients to receive either CBD dominant or placebo, and follow them for six months to confirm our ability to recruit patients, adhere to protocol, and capture full outcome data for at least 85% of patients.

DETAILED DESCRIPTION:
Approximately 25% of patients develop persistent post-surgical pain (PPSP) after undergoing total knee arthroplasty (TKA), and higher pre-surgery and acute post-operative pain are associated with this outcome. Medicinal cannabis has anti-inflammatory and analgesic properties and may reduce peri-operative pain and the rate of PPSP following TKA. Cannabidiol (CBD) is the active ingredient of interest because of its anti-inflammatory effects and lack of psychoactive effects seen with tetrahydrocannabinol (THC). The primary objective of this pilot trial is to assess the feasibility of a definitive trial to determine the effect of medicinal cannabis, versus placebo, on the proportion of patients experiencing PPSP following TKA. The primary objective of the definitive trial is to determine if medicinal cannabis add-on therapy, versus placebo, reduces the proportion of patients experiencing PPSP at 6 months following TKA. The secondary objectives of the definitive trial are to determine if medicinal cannabis, versus placebo, reduces opioid use, reduces peri-operative pain interference, improves physical functioning, mental functioning, return to function, anxiety and depression, and sleep. The effect of medicinal cannabis, versus placebo, on the incidence of adverse events at 6 months post-surgery will also be examined. In this blinded multi-centre pilot trial, 40 patients will be randomized to receive either oral capsules of CBD oil or visually identical placebo in addition to standard of care pain medications. Participants will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TKA aged 18 or older
* Cognitive ability and English-language skills required to complete outcome measures
* Provision of informed consent
* Successful completion of the run-in period

Exclusion Criteria:

* Severe cardio-respiratory disease (For operationalizing: ASA 4/NYHA 4)
* Substance use disorder based on DSM-V criteria
* Allergy or intolerance to cannabis, cannabis derivatives, or other ingredients of the study drug
* Patients who are pregnant, planning to be pregnant, or breastfeeding
* Revision TKA
* Bilateral TKA
* Presenting for their pre-surgical consultation less than 4 weeks before surgery
* Patients with a chronic pain condition affecting the knee (other than osteoarthritis) (e.g.: patients with knee pain due to fibromyalgia or chronic pain syndrome will be excluded)
* Unwilling or unable to follow the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Persistent post-surgical pain (PPSP) | 6 months
  Proportion of patients experiencing moderate to severe PPSP (average of pain over last week of ≥4 out of 10 on a numeric rating scale [NRS])

SECONDARY OUTCOMES:
Opioid use | 6 months
  Use of opioids (mean morphine equivalent dose [MED] change)
Peri-operative pain intensity | 24-48 hours, 2-weeks, 6-weeks, 3-months and 6-months
  Peri-operative pain measured on an 11-point NRS
Pain interference | 24-48 hours, 2-weeks, 6-weeks, 3-months and 6-months
  Pain interference measured by the Brief Pain Inventory (BPI-SF)
Physical function | 6 months
  Physical component summary (PCS) score of the SF-12
Mental function | 6 months
  Mental component summary (MCS) score of the SF-12
Return to function | 6 months
  Return to 80% of pre-injury function (work, leisure, home activities)
Insomnia | 6 months
  Insomnia symptoms on the Insomnia Severity Index (ISI)
Anxiety and depression | 6 months
  Anxiety and depression on the Hospital Anxiety and Depression Scale (HADS)
Safety - Adverse events | 6 months
  Serious and non-serious adverse events

OTHER OUTCOMES:
Feasibility - recruitment | 6 months
  Ability to recruit 40 patients
Feasibility - retention | 6 months
  Ability to follow 85% of patients
Feasibility - compliance | 6 months
  Patient compliance with the study treatment (75% of patients comply with 75% of the study doses)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Adili, MD, P.Eng, Principal Investigator — McMaster University; Jason W Busse, DC, PhD, Principal Investigator — McMaster University; Vahid Ashoorion, MD, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided